CLINICAL TRIAL: NCT03141593
Title: Oral Vitamin D Substitution Weekly or Monthly - Which Procedure Leads to Highest Adherence? A Prospective Intervention Study in Outpatient Care
Brief Title: Oral Vitamin D Substitution Weekly or Monthly and Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00300
Record Dates: First submitted 2017-03-23; First posted 2017-05-05 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Vitamin D Deficiency
Keywords: adherence to medication; electronic monitoring
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Patient will be recruited by their general practitioners (GP) and allocated to the GP's form (liquid or solid). Patients will be randomly assigned to start weekly or monthly intake for 3 months, and switch to the other frequence for 3 more months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D: liquid form, start weekly (Active Comparator): 5'600 IU weekly (1.4 ml oily drops) start for 3 months, will cross-over to 24'000 IU monthly (5 ml alcoholic drops) for the following 3 months.
  Interventions: Drug: Vitamin D: liquid form, start weekly
- Vitamin D: solid form, start weekly (Active Comparator): 5'600 IU weekly (1 soft capsule) start for 3 months, will cross-over to 20'000 IU monthly (1 tablet) for the following 3 months.
  Interventions: Drug: Vitamin D: solid form, start weekly
- Vitamin D: liquid form, start monthly (Active Comparator): 24'000 IU monthly (5 ml alcoholic drops) start for 3 months, will cross-over to 5'600 IU weekly (1.4 ml oily drops) for the following 3 months.
  Interventions: Drug: Vitamin D: liquid form, start monthly
- Vitamin D: solid form, start monthly (Active Comparator): 20'000 IU monthly (1 tablet) start for 3 months, will cross-over to 5'600 IU weekly (1 soft capsule) for the following 3 months.
  Interventions: Drug: Vitamin D: solid form, start monthly

INTERVENTIONS:
Drug: Vitamin D: liquid form, start weekly — Patient will start treatment with weekly schedule, and switch after 3 months to monthly schedule for another 3 months.
  Other Names: Vitamin D3 Streuli
  Arms: Vitamin D: liquid form, start weekly
Drug: Vitamin D: liquid form, start monthly — Patient will start treatment with monthly schedule, and switch after 3 months to weekly schedule for another 3 months.
  Other Names: Vi-De 3 Monatsdosis
  Arms: Vitamin D: liquid form, start monthly
Drug: Vitamin D: solid form, start weekly — Patient will start treatment with weekly schedule, and switch after 3 months to monthly schedule for another 3 months.
  Other Names: Dekristolvit D3
  Arms: Vitamin D: solid form, start weekly
Drug: Vitamin D: solid form, start monthly — Patient will start treatment with monthly schedule, and switch after 3 months to weekly schedule for another 3 months.
  Other Names: Dekristol
  Arms: Vitamin D: solid form, start monthly

SUMMARY:
Vitamin D deficiency (defined as 25(OH)-vitamin D serum level <50 nmol/l) is cured with supplementation by mouth. National guidelines recommend the administration of 800 IU cholecalciferol daily for an effective treatment, especially during the winter (poor sun exposition). Commercially available pharmaceutical forms are liquid in Switzerland (drops) and solid forms in Germany (tablets and capsules). Because therapeutic range of vitamin D3 is wide and toxicity is seldom reached, even after the consumption of 200'000 IU, and because the administration of 8 drops daily is inconvenient, weekly and monthly administrations of the cumulative amount (i.e., 5'600 IU weekly or 24'000 IU monthly) have been investigated. Both administration schedules are therapeutic equivalent. The study aims to investigate which form (liquid or solid) and which schedule (weekly or monthly) procure the highest adherence behavior with outpatients under polypharmacy i.e., with 4 or more medications daily. The investigators will use commercially available Swiss and German products.

DETAILED DESCRIPTION:
Intervention study in patients with serum vitamin D <50 nmol/l and polypharmacy, defined as ≥4 medicaments/day. Treatment duration: 6 months. Treatment groups are defined as Lm (liquid monthly 24'000 IU); Lw (liquid weekly 5'600 IU); Sm (solid monthly 20'000 IU) and Sw (solid weekly 5'600 IU). Cross-over design with identical form (liquid or solid) and switching frequence, i.e. from weekly to monthly treatment and vice versa, for 3 months each.

ELIGIBILITY:
Inclusion Criteria:

* vitamin D deficiency by serum level <50 nmol/l
* polypharmacy defined as 4 daily medicines or more
* speaking German or Swiss German

Exclusion Criteria:

* hypercalcaemia
* substitution treatment with cholecalciferol in the past 3 months
* medication intake provided by a third person and not by the patient himself

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Adherence to medication | 3 months of treatment
  Taking adherence: number of dosis taken divided by number of dosis prescribed. Timing adherence: number of dosis taken within a time interval (within 15% of the mean preset intake time) divided by number of dosis prescribed.

SECONDARY OUTCOMES:
Serum level of vitamin D | 3 and 6 months
  Level of serum vitamin D compared to baseline value.
Patients preferences | 3 months of treatment
  Questionnaire with 5-point Likert scale (from 1=strongly disagree to 5=strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Prof, Study Director — University of Basel
Locations (1):
- Pharmaceutical Care Research Group, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
not decided yet